CLINICAL TRIAL: NCT05079880
Title: Effect of Caffeine on Time to Anesthetic Emergence After Laparoscopic Cholecystectomy : Randomized-controlled Trial
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tunis University (Other)
Responsible Party: Principal Investigator, Daghmouri Mohamed Aziz, Principal investigator, Tunis University
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: HTHEC-2017-09
Record Dates: First submitted 2021-09-21; First posted 2021-10-15 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Laparoscopic Cholecystectomy
Keywords: Caffeine; Anesthesia emergence; Cholecystectomy; Sevoflurane

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GC group (Experimental): received 300 mg of caffeine citrate infusion
  Interventions: Drug: 300 mg of caffeine citrate infusion
- GS group (Placebo Comparator): Equivalent saline infusion
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 300 mg of caffeine citrate infusion — At the end of the surgery, the study drug was given intravenously over ten minutes than the sevoflurane infusion was stopped corresponding to the start of the recovery period
  Arms: GC group
Drug: Placebo — At the end of the surgery, the placebo was given intravenously over ten minutes than the sevoflurane infusion was stopped corresponding to the start of the recovery period
  Arms: GS group

SUMMARY:
A faster emergence from general anesthesia has a double medico-economic impact by reducing the risks of complications and optimizing the performance of surgical units. No drug has been retained for its ability to actively accelerate anesthetic emergence by antagonizing hypnotics. Thus, the aim of this study was to examine the effect of caffeine on the time to emerge from sevoflurane anesthesia for laparoscopic cholecystectomy.

ELIGIBILITY:
Inclusion Criteria:

* American society of Anesthesiologists (ASA) I and II patients, aged older than 18 years old and scheduled for laparoscopic cholecystectomy

Exclusion Criteria:

* Patient with an allergy to caffeine citrate and analgesics used during postoperative period, those with severe renal or hepatic failure, those who refused to participate in addition to patient with heart rhythm disorder, seizure disorder, hypertension, alcoholic or psychiatric illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-08-15 (Actual); Primary Completion 2021-10-15 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
anesthetic recovery time | Postoperative
  time to return to spontaneous breathing, eye opening on verbal command and time for extubation

SECONDARY OUTCOMES:
plasma caffeine levels at H1 and H24 | Hour 1 and Hour 24
postoperative rehabilitation | 24 hours postoperatively
  incidence of headache, nausea and vomiting, tiredness score, time to the first flatus and satisfaction of patients
postoperative pain (Visual Analog Scale score 0 "no pain" to 10 "severe pain") and consumption of morphine | 24 hours postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Habib Thameur Hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided